CLINICAL TRIAL: NCT05468723
Title: Evaluating Patient Comfort and Environmental Conditions in the Carecube Negative Pressure Isolation Chamber.1
Status: Completed | Type: Observational
Sponsor: Carecubes, Inc. (Industry)
Collaborators: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: TP-00003 Revision: 05
Record Dates: First submitted 2022-07-18; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Infectious Diseases
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Carecube Negative Pressure Isolation Chamber — Subjects will be tasked to stay within the Carecube Isolation Chamber for at least 4 hours and have 3 consecutive timepoints illustrating a plateau level for all participants parameters. Environmental data will be collected by physicians and nurses [which may include physicians, physician assistants, Registered Nurses, Licensed Practical Nurses, medical technicians and emergency medical technicians (EMTs)] . Additionally, atmospheric Oxygen, Carbon Dioxide, humidity, and room temperature will be monitored and recorded on an hourly basis. External to the room humidity and temperatures will also be recorded. The participant will be exposed to room temperature (° Fahrenheit) and humidity (RH%), ranging from 65°- 90° Fahrenheit and 30%-60% RH. Participants will also be asked to record on a questionnaire, in order to demonstrate that the Carecube Negative Pressure Isolation chamber is a safe and non-hostile environment for the patients that will be contained during normal operations.

SUMMARY:
This is a human non-significant risk (NSR) clinical study designed to objectively and participatively verify that the Carecube Negative Pressure Isolation Chamber is a safe and non-hostile environment for the patients that will be contained within the chamber during normal operations.

DETAILED DESCRIPTION:
Device Information:

The Carecube Negative Pressure Isolation Chamber is a patient isolation unit (PIU) designed for the temporary isolation of patients within a hospital to prevent particulate (biological) cross-contamination between user and patient, while enclosing the contaminated patient from the external environment.

Study Description:

Participants will be tasked to stay within the Carecube Negative Pressure Isolation Chamber for a minimum of three consecutive time points (1 hour apart) illustrating a plateau level for all parameters, up to a maximum of 7 hours (readings will be taken at baseline and hourly thereafter).

The Carecube Negative Pressure Isolation Chamber will be set up indoors, in an emergency department and hospital floor environment. We will collect data and demonstrate that the Carecube Isolation chamber is a safe and non-hostile environment for the patients that will be contained within, during normal operations.

Each participant will be asked to come to a test center facility to complete and sign the informed consent and receive instruction to interact with the simulation. Subjects will be tasked to stay within the Carecube Isolation Chamber for at least 4 hours and have 3 consecutive timepoints illustrating a plateau level for all participants parameters.

Environmental data will be collected by physicians and nurses. Additionally, atmospheric Oxygen, Carbon Dioxide, humidity, and room temperature will be monitored and recorded. External to the room humidity and temperatures will also be recorded. The participant will be exposed to room temperature (° Fahrenheit) and humidity (RH%), ranging from 65°- 90° Fahrenheit and 30%-60% RH. Participants will also be asked to record on a questionnaire, in order to demonstrate that the Carecube Negative Pressure Isolation chamber is a safe and non-hostile environment for the patients that will be contained during normal operations.

ELIGIBILITY:
Inclusion Criteria:

Male, female, non-binary between the ages of 19-65 No existing medical condition that would impact the Subject from staying within the containment system for the specified time-period.

Patient is not pre-dispositioned for claustrophobia

Exclusion Criteria:

Subjects that have a pre-existing condition of claustrophobia Subjects that have a history of hypertension Subjects with a clinical diagnosis of generalized anxiety disorder (GAD) Subjects with a clinical diagnosis of major depressive disorder (MDD) Morbidly obese patients (BMI above 40) Subjects who are Women of Child Bearing Potential (WOCBP) who either are pregnant or suspect they are pregnant

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community members
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2022-06-18 (Actual); Study Completion 2022-06-18 (Actual)

PRIMARY OUTCOMES:
Body Temperature | 4 hours
  Subject's body temperature maintains a normal healthy value based on their entry body temperature and outside the Carecube
Blood Pressure | 4 hours
  Subject's blood pressure stays at a normal healthy level with respect to their initial baseline
Pulse | 4 hours
  Subject's pulse stays within a normal healthy level based with respect to their initial baseline
Oxygen levels | 4 hours
  Subject's Oxygen levels stays within a normal healthy level based with respect to their initial baseline
Movement | 4 hours
  Subject is able to move within the Carecube, to include activities such as sitting up, laying down, rotating, foot flexion or other body positioning within the hospital bed located within the Carecube.
Communication | 4 hours
  Subject and provider are able to clearly and effectively communicate while the Subject is positioned within the Carecube Negative Pressure Isolation Chamber.
Environmental Condition | 4 hours
  Environment does not have an elevation of temperature, Carbon Dioxide and humidity outside a normal range as compared to the external environment of the chamber.

SECONDARY OUTCOMES:
Comfort | 4 hours
  Subject does not become uncomfortable or claustrophobic
Anxiety | 4 hours
  Subject does not become anxious

CONTACTS AND LOCATIONS:
Overall Officials: Andy Schnaubelt, Principal Investigator — UNMC
Locations (1):
- UNMC, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Undecided